CLINICAL TRIAL: NCT07161921
Title: Integrative Metagenomic and Metabolomic Profiling Identifies Gut Microbiota and Metabolite Signatures Associated With Lymph Node Metastasis in Pancreatic Cancer
Brief Title: Gut Microbiota and Metabolite Signatures Associated With Lymph Node Metastasis in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-PCAMICROBE-3
Record Dates: First submitted 2025-06-04; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer; Microbial Colonization; Lymph Node Metastasis
Keywords: pancreatic cancer; microbiome; metabolite; lymph node metastasis
MeSH Terms: conditions — Pancreatic Neoplasms; Communicable Diseases; Lymphatic Metastasis | interventions — lncRNA LNMAT1, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — metagenomics of microbiome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lymph node metastasis: Histopathological examination confirmed the presence of at least one lymph node metastasis
  Interventions: Other: lymph node metastasis
- non-lymph node metastasis: Histopathological examination confirmed the absence of at least one lymph node metastasis

INTERVENTIONS:
Other: lymph node metastasis — Histopathological examination confirmed the presence of at least one lymph node metastasis
  Groups: lymph node metastasis

SUMMARY:
This study investigates the association between gut microbiota and lymph node metastasis (LNM) in pancreatic cancer. While gut microbial dysbiosis has been linked to pancreatic cancer development and distant metastasis, its role in LNM remains unclear. By comparing the gut microbiota and metabolite profiles of patients with and without LNM, the study aims to identify key microbial and metabolic signatures linked to metastasis. Additionally, predictive models will be developed to facilitate preoperative identification of high-risk patients, with the goal of improving clinical decision-making and treatment planning.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most aggressive malignancies of the digestive system, characterized by an insidious onset, early lymph node metastasis (LNM), poor prognosis, and resistance to chemotherapy and radiotherapy. LNM is recognized as an independent prognostic factor affecting patient survival.

Dysbiosis of the gut microbiota has been implicated in cancer development and progression by influencing metabolic and immune functions. Previous studies demonstrated that gut microbiota is altered in patients with pancreatic cancer, and microbial signatures may serve as potential diagnostic markers. Moreover, gut microbiota has been reported to predict distant metastasis in pancreatic cancer patients. However, the relationship between gut microbiota and lymph node metastasis in pancreatic cancer remains unexplored.

This study aims to characterize the differences in gut microbial composition between pancreatic cancer patients with and without LNM, identify key microbial taxa and metabolites associated with LNM, and elucidate their potential roles in mediating metastasis. Furthermore, we seek to develop predictive models based on microbiome and metabolite profiles for LNM to facilitate preoperative identification of high-risk patients, ultimately optimizing clinical decision-making and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Agree to participate in the study

Exclusion Criteria:

* A prior diagnosis of other malignancies, infectious diseases, psychiatric or neurodegenerative disorders, or conditions affecting the oral or gastrointestinal systems;
* Recent medical treatments or procedures within specific time frames, including: (a) Use of antibiotics, hormone therapy, or immunosuppressive agents within the past three months. (b) Undergoing gastrointestinal reconstructive surgery within the past three months. (c) Regular use of laxatives, antidiarrheal medications, or high-dose probiotics within the past month. (d) Participation in gastrointestinal examinations within the past three days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pancreatic cancer and received radical surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
microbiota profiles | Through the completion of study, an average of 3 years
  microbiota profile by metagenomic of the two groups

SECONDARY OUTCOMES:
metabolite profiles | Through the completion of study, an average of 3 years
  metabolite profile by metabolomic of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, Professor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
metagenomics and metabolites data are to be shared with other researchers